CLINICAL TRIAL: NCT00370721
Title: Intravitreal Bevacizumab for Management of Active Progressive Proliferative Diabetic Retinopathy (PDR)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8538
Record Dates: First submitted 2006-08-30; First posted 2006-09-01 (Estimated); Last update posted 2008-06-26 (Estimated); Status verified 2008-06

CONDITIONS: Diabetic Retinopathy
Keywords: Proliferative diabetic retinopathy(PDR); Pan retinal photocoagulation (PRP); Vitreous hemorrhage; Traction retinal detachment; Neovascularization on disc (NVD); Neovascularization elsewhere (NVE); Fibrous proliferation on disc (FPD); Fibrous proliferaiton elsewhere (FPE)
MeSH Terms: conditions — Diabetic Retinopathy; Vitreous Hemorrhage | interventions — Bevacizumab

ARMS (1):
- I (Experimental)
  Interventions: Drug: bevacizumab

INTERVENTIONS:
Drug: bevacizumab

SUMMARY:
To evaluate the effect of intravitreal bevacizumab on the course of diabetic retinopathy in cases with the signs of active progressive PDR

ELIGIBILITY:
Inclusion Criteria:

* Cases of active progressive PDR with history of scatter laser photocoagulation

Exclusion Criteria:

* history of vitrectomy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2006-03

PRIMARY OUTCOMES:
Regression of diabetic retinopathy
visual acuity

SECONDARY OUTCOMES:
neovascularization
fibrous proliferation
traction retinal detachment
vitreous hemorrhage
pan retinal photocoagulation

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Ahmadieh, MD, Principal Investigator — Ophthalmic Research Center of Shaheed Beheshti Medical University
Locations (1):
- Hamid Ahmadieh, MD, Tehran, Tehran Province, Iran